CLINICAL TRIAL: NCT00203138
Title: A Multicenter, Open-Label, Phase III Study for the Safety, Tolerability and Clinical Effect of Rasagiline Mesylate in Patients With Parkinson's Disease
Brief Title: Safety, Tolerability, and Effectiveness of Rasagiline Mesylate in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Siyu Liu, MD, VP, Global Head Clinical Operations, Teva Branded Pharmaceutical Products
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVP - 1012/233
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

INTERVENTIONS:
Drug: rasagiline mesylate

SUMMARY:
Patients who completed the study TVP-1012/232 are eligible to enter the extension study to continue their rasagiline therapy for their Parkinson's disease (PD). During this study the patient's safety, tolerability of rasagiline, and effectiveness of this therapy will be monitored.

ELIGIBILITY:
Inclusion Criteria:

• Patients who completed evaluations of week 52 of the TVP 1012/232 protocol, where continued rasagiline therapy is warranted, in the opinion of the principal investigator

Exclusion Criteria:

• Patients having suffered adverse effects that were probably drug-related in the TVP-1012/232 study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2004-06; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Tolerability - Number of patients completing study on their original treatment assignment (dose reduction and dropout) | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Salzman, Ph.D., Study Director — Teva Neuroscience, Inc.